CLINICAL TRIAL: NCT05420610
Title: Early Goal-Directed Therapy Utilizing Transpulmonary Thermodilution for Treating Adult Patients With Severe Burn Injury
Brief Title: Early Goal-Directed Therapy Utilizing Transpulmonary Thermodilution and Severe Burn Injury
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101364B0
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with major burn.: Adult patients (age > 18 years) suffered from major burn which defined as total burned surface area (TBSA) > 20% with at least second degree burn depth were admitted to the intensive care unit (ICU) of the Burn Center at a tertiary medical center were retrospectively reviewed.
  Interventions: Other: Control group: Patients being admitted when The advancement of transpulmonary thermodilution(TPTD) device was unavailable.; Other: Study group: TPTD device was implemented for monitoring.

INTERVENTIONS:
Other: Control group: Patients being admitted when The advancement of transpulmonary thermodilution(TPTD) device was unavailable. — The control group included patients being admitted when TPTD device was unavailable; and relatively stable patients without the need for TPTD. The adequacy of fluid resuscitation in the control group was monitored by traditional monitoring parameters including vital signs and hourly urine output.
Other: Study group: TPTD device was implemented for monitoring. — TPTD device was implemented for monitoring; the inclusion criteria included patients suffering from 2nd degree burn greater than 40% TBSA; a combined 2nd to 3rd degree burn greater than 30% TBSA; or patients with inhalation injury despite the burned surface area.

SUMMARY:
This study aimed to optimize fluid resuscitation with transpulmonary thermodilution (TPTD)-guided protocol and to lower the mortality rate of the severely burned.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years).
* Major burn (as total burned surface area (TBSA) > 20% with at least second degree burn depth).
* Admitted to the intensive care unit (ICU) of the Burn Center.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with severe cardiopulmonary diseases, or associated with other major trauma.
* Patient with incomplete data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2011 to June 2019, all adult patients (age > 18 years) suffered from major burn,23 defined as total burned surface area (TBSA) > 20% with at least second degree burn depth were admitted to the intensive care unit (ICU) of the Burn Center at a tertiary medical center were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Patient mortality | Up to 6 months
  The primary outcome was patient mortality after major burn.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan